CLINICAL TRIAL: NCT04718636
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 2-WAY CROSSOVER STUDY ON THE EFFECTS OF CC-99677 ON THE PHARMACOKINETICS OF AN ORAL CONTRACEPTIVE IN HEALTHY FEMALE SUBJECTS
Brief Title: A Study to Evaluate Effects of CC-99677 on the Pharmacokinetics of an Oral Contraceptive in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-99677-CP-003; U1111-1258-2701 (Registry Identifier: WHO)
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Female Volunteers; CC-99677; Contraceptive
MeSH Terms: interventions — Contraceptives, Oral; norgestimate, ethinyl estradiol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of OC alone, then progress to OC in combination with CC-99677 (Experimental): Oral Contraceptive (OC) and CC-99677 will be administered daily
  Interventions: Drug: Oral Contraceptive (Ortho Tri-Cyclen or its generic equivalent); Drug: CC-99677

INTERVENTIONS:
Drug: Oral Contraceptive (Ortho Tri-Cyclen or its generic equivalent) — Daily
Drug: CC-99677 — Daily

SUMMARY:
The purpose of this study is to evaluate the effect of CC-99677 coadministration on the pharmacokinetics (PK) of an oral contraceptive (OC).

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following criteria to be eligible for enrollment into the study:

1. Participant is ≥ 18 and ≤ 48 years of age at the time of signing the informed consent form (ICF).
2. Participant must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Participant is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Participant is in good health, as determined by the Investigator based on a physical examination at screening.
5. Participant has a body mass index (BMI = weight [kg]/(height [m])2) between 18 and 30 kg/m2 (inclusive).
6. Females of childbearing potential (FCBP) must have a negative pregnancy test at screening and baseline as verified by the Investigator prior to the first dose of IP. She must agree to ongoing pregnancy testing during the course of the study, and prior to discharge from the study site. This applies even if the FCBP participant practices true abstinence from heterosexual contact.
7. FCBP must either commit to true abstinence from heterosexual contact (which must be reviewed on a weekly basis, as applicable, and source documented) or agree to use, and be able to comply with, highly effective methods of contraception without interruption, during the study (including any dose interruptions), and for at least 28 days after discontinuation of IP.
8. If previously taking a hormonal OC, she must agree to continue using (or switch over to, if applicable) Ortho Tri-Cyclen® or its generic equivalent, which is to be provided by the study center, throughout the study.
9. Female participants NOT of childbearing potential must:

   • Have been surgically sterilized (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy; proper documentation is required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle stimulating hormone [FSH] level of > 40 IU/L at screening).
10. Participant has clinical laboratory safety test results that are within normal limits or considered not clinically significant by the Investigator. In addition, ALT, AST, and total bilirubin must be less than the upper limit of normal at screening and on Day -1.
11. Participant is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
12. Participant has normal or clinically acceptable 12 lead ECG with a QTcF value ≤ 450 msec at screening.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Participant has any significant medical condition (including but not limited to gynecologic, infectious, oncologic, neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders), laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
2. Participant has any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study according to the Investigator or Sponsor.
3. Participant has any condition that confounds the ability to interpret data from the study.
4. Pregnant, breast-feeding, or < 6 months postpartum at the time of ICF signing.
5. Any condition that contraindicates the use of OCs.
6. History of irregular menses, pregnancy, or adverse experiences while taking OCs.
7. Use of hormonal contraceptives other than OCs (eg, transdermal patch, vaginal ring, intrauterine device) within 3 months, implanted contraceptives within 6 months, or injectable contraceptives for 12 months prior to screening.
8. History of two or more drug allergies.
9. History of allergy to Ortho Tri-Cyclen® or its generic equivalents.
10. Presence of any clinically significant allergic disease (excluding non-active seasonal allergies like hay fever). Participant was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
11. Participant has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days prior to the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer). Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
12. Participant has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration. Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
13. Participant has used CYP3A inducers and/or inhibitors (including St. John's Wort) within 30 days preceding the first dose administration.
14. Participant has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, or excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable. Other previous surgeries may be acceptable with concurrence of the Sponsor's Medical Monitor.
15. Participant donated blood or serum within 8 weeks before the first dose administration to a blood bank or blood donation center.
16. Participant has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual or other country-specific guideline within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
17. Participant has a history of alcohol abuse or other country-specific guideline within 2 years before the first dose administration, or positive alcohol screen.
18. Participant is known to have a history of hepatitis B and/or hepatitis C, or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.

    a. Note: Participants who received hepatitis B vaccination and who test positive for hepatitis B surface antibody and negative for both hepatitis B surface antigen and hepatitis B core antibody remain eligible for study participation.
19. Participant is older than 35 years of age and smokes any number of cigarettes per day or the equivalent in other tobacco products (self-reported).
20. Participant is 35 years of age or younger and smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
21. Participant has a history of incompletely treated Mycobacterium tuberculosis (TB) infection, as indicated by:

    1. Participant's medical records documenting incomplete treatment for Mycobacterium TB
    2. Participant's self-reported history of incomplete treatment for Mycobacterium TB
    3. Note: Participants with a history of TB who have undergone treatment accepted by the local health authorities (documented) may be eligible for study entry
22. Participant has received immunization with a live or live attenuated vaccine within 2 months prior to the first dose administration or is planning to receive immunization with a live or live attenuated vaccine for 2 months following the last dose administration.
23. Participant has a history of Gilbert's syndrome or has laboratory findings at screening that, in the opinion of the Investigator, are indicative of Gilbert's syndrome.
24. Participants with clinical symptoms or signs suggesting active, subacute, or unresolved chronic infection. All questions regarding this criterion should be discussed with the Sponsor.
25. Participant has previously been exposed to CC-99677 (eg, in a prior clinical trial).
26. Participant has a history of photosensitivity to medications.
27. Participant is part of the study site staff personnel or a family member of the study site staff.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - AUC0-τ | Up to 36 hours post-dose
  The area under the curve (AUC) for the defined interval between doses (TAU)
Pharmacokinetic - AUC0-t | Up to 36 hours post-dose
  The area under the curve (AUC) from the time of dosing to the last measurable concentration
Pharmacokinetic - Cmax | Up to 36 hours post-dose
  Maximum observed plasma concentration occurring at Tmax
Pharmacokinetic - Tmax | Up to 36 hours post-dose
  The time of maximum observed concentration sampled during a dosing interval
Pharmacokinetic - t1/2 | Up to 36 hours post-dose
  Terminal half-life
Pharmacokinetic - CL/F | Up to 36 hours post-dose
  The total body clearance for extravascular administration divided by the fraction of dose absorbed, calculated using the observed value of the last non-zero concentration
Pharmacokinetic - Vz/F | Up to 36 hours post-dose
  The volume of distribution associated with the terminal slope following extravascular administration divided by the fraction of dose absorbed, calculated using the observed value of the last non-zero concentration

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Kofi Mensah, MD, PhD, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Qps-Mra, Llc, Miami, Florida
  - Hassman Research Institute, Marlton, New Jersey
  - PPD Phase 1 Clinic, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/